CLINICAL TRIAL: NCT04595877
Title: Double-blind, Randomized Controlled Study to Assess the Analgesic Effect of a Single Intravenous Dose of 2 g of Magnesium Dipyrone (Metamizol) and Changes in Plasma Beta-endorphin Immunoreactivity (Beta-EPIr) Values in Patients Undergoing Elective Inguinal Herniorrhaphy (Bassini Operation) Under Epidural Anesthesia.
Brief Title: Double-blind, Randomized Controlled Study to Assess the Analgesic Effect of 2 g of Magnesium Dipyrone (Metamizol) and Changes in Plasma Beta-endorphin Immunoreactivity Values in Patients Undergoing Elective Inguinal Herniorrhaphy Under Epidural Anesthesia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonio Martín Duce (Other)
Responsible Party: Sponsor-Investigator, Antonio Martín Duce, Dr. Antonio Martin Duce, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1093-10
Record Dates: First submitted 2020-09-23; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Pain; Beta-endorphin; Dipyrone; Hernia Surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts will be kept blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dipyrone group (Experimental): Dipyrone 2 g (Nolotil®, Europharma, Madrid, Spain); one ampoule in 50 mL of 0.9% saline solution as an intravenous infusion over 10 min.
  Interventions: Drug: Dipyrone administration; Behavioral: Pain assessment; Biological: beta-endorphin immunoreactivity
- Placebo group (Placebo Comparator): The placebo will be matched to the study drug for, color, and size. Placebo will be administered in a single dose in 50 mL of 0.9% saline solution as an intravenous infusion over 10 min.
  Interventions: Behavioral: Pain assessment; Biological: beta-endorphin immunoreactivity; Other: Placebo administration

INTERVENTIONS:
Drug: Dipyrone administration — Dipyrone 2 g (Nolotil®, Europharma, Madrid, Spain); one ampoule in 50 mL of 0.9% saline solution as an intravenous infusion over 10 min.
  Arms: Dipyrone group
Behavioral: Pain assessment — Pain will be evaluated by the patient according to a 100-mm visual analogue scale (VAS) (from point 0 "no pain" to point 10 "unbearable pain").
Biological: beta-endorphin immunoreactivity — Plasma beta-EPIr levels will be measured by an immunoradiometric assay (Allegro Beta-endorphin, Nichols Institute Diagnostics, SAN JUAN DE CAPISTRANO, CA) (normal values 29-40 pg/mL). It will be obtained by venous blood samples (5 mL) at the same time points at pain will be measured.
Other: Placebo administration — Placebo in 50 mL of 0.9% saline solution as an intravenous infusion over 10 min.
  Arms: Placebo group

SUMMARY:
A double-blind, randomized controlled study is designed to assess the analgesic effect of a single intravenous dose of 2 g of magnesium dipyrone (metamizol) and whether the administration of the active drug will be associated with changes in plasma beta-endorphin immunoreactivity values in patients undergoing elective inguinal herniorrhaphy (Bassini operation) under epidural anesthesia. Participants, care givers, and those assessing the outcomes will be blinded to group assignment. Participants will be randomized to receive dipyrone or a placebo. The active drug or placebo will be administered as an intravenous infusion over 10 min. Pain will be evaluated by the patient according to a 100-mm visual analogue scale. Assessments will be carried out the day before surgery, immediately after operation, at the time of drug administration, and 60 and 180 min after treatment. At the same time as pain will be evaluated, blood samples will be drawn for plasma beta-endorphin immunoreactivity measurement (immunoradiometric assay).

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years, elective surgery, routine laboratory tests (blood cell count, biochemical profile, urinalysis), chest radiography, twelve-lead electrocardiography, body mass index (BMI), blood pressure, pulse rate normal or abnormal values without clinical relevance and a mental status sufficient to be able to complete efficacy tests.

Exclusion Criteria:

* Patients who had taken other analgesics or anti-inflammatory drugs 24 h before surgery, as those with known hypersensitivity to the drug or with any other disorder contradicting the administration of dipyrone. Patients with hypersensitivity to non-steroidal anti-inflammatory agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Analgesic efficacy-Pain relief | 30 seconds
  Visual Analogue Scale score

SECONDARY OUTCOMES:
Beta-endorphins levels. | 1 minute
  Beta-endorphin immunoreactivity levels

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing and Physiotherapy Department, Madrid, Alcalá de Henares, Spain

IPD SHARING:
Plan to Share IPD: No